CLINICAL TRIAL: NCT03231020
Title: Parental Experience in the Single Ventricle Interstage Utilizing a mHealth Innovation: A Comparative Case Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: American Nurse Credentialing Center (Unknown)
Responsible Party: Principal Investigator, Lori Erickson, CHAMP Clinical Program Manager, MSN, CPNP-PC, Children's Mercy Hospital Kansas City
Other Study IDs: 17050339
Record Dates: First submitted 2017-07-12; First posted 2017-07-27 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: mHealth; Adherence, Patient
Keywords: single ventricle; pediatric cardiology; interstage; home monitoring; mHealth
MeSH Terms: conditions — Patient Compliance; Univentricular Heart | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adherent Group: Parent(s) that submitted a high rate of data transfer (top 25th percentile) with rate of data days of mHealth technology for data transfer
  Interventions: Other: Interview
- Non-Adherent Group: Parent(s) that chose to return mHealth technology before the end of the interstage period and/or low rate of data transfer (bottom 25th percentile) with rate of data days
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — The proposed research study uses a comparative case study methodology, utilizing multiple sources of data to deeply examine 8-10 "cases," each of which is defined as parent(s) of a child (< 5 years of age) with single ventricle disease who used the mHealth application. One group of cases (4-5) will have used the mHealth application less than recommended (non-adherent to the home monitoring recommendations) or declined to use the application and returned it before the end of the interstage period. The other group of comparison cases (4-5 cases) will have used the application as recommended by the clinical team (adherent) and continued doing so through the interstage period.

SUMMARY:
The purpose of this study is to provide a rich description of the parental perspectives of utilizing a mHealth application for data transfer during the single ventricle interstage monitoring period. A gap in the body of knowledge of single ventricle cardiac disease interstage will be explored with these research questions: 1) How do parents of children (< 5 years of age) with single ventricle disease describe their experiences using a mHealth application during the interstage period (first 6-12 months of child's life)? And 2) How do these experiences influence their decision making for use of the mHealth application?

DETAILED DESCRIPTION:
Background Nearly 2,000 infants with single ventricle cardiac disease are born each year in the United States, and have near certain mortality without surgical intervention. The heart with this congenital disease can never be converted to a four-chambered heart but rather, a palliative three-staged surgical strategy has been designed to maintain both circulation to the body and lungs without a pump. After an initial neonatal surgery, most infants are discharged home and return for a second surgery around six months of life. The time occurring between surgeries is known as the interstage period. This interstage period is very high risk and high demand time for parents, and there is a mortality rate during the interstage ranging from 2-20%, often from unknown reasons.

Hypoplastic left heart syndrome (HLHS) is a specific type of single ventricle disease that is one of the most complex forms of congenital heart disease. Publications have focused on improving the care of infants with HLHS using a Quality Improvement Model with the National Pediatric Cardiology Quality Improvement Collaborative (NPCQIC) through reduced variation, best practices, and transparency. The concept of interstage home monitoring to reduce mortality also was primarily focused on infants with only HLHS until recently when the focus was made onto comprehensive care from birth to 1 year of age. Hemodynamic data such as oxygen saturation, heart rate, intake, and overall status from a parental perspective were used to promote communication and attempts of early recognition of deterioration in this high-risk population. A strong set of qualitative studies have come from Rempel et al. in Canada on a cross-section of mainly white married parents of infants with HLHS and their parenting experience. Parenting under Pressure and the Facets of parenting a child with HLHS were studies which used the grounded theory approach and provided substantial additions to our knowledge of the interstage HLHS parenting experience. The basis of much of the care for all types of single ventricle cardiac disease at home is found from the care of HLHS and applied to infants with all types of single ventricle anatomy.

Most hospitals with pediatric cardiac surgery programs have interstage home monitoring programs for high risk infants with single ventricle heart disease to provide care and support for infants with all types of single ventricle cardiac disease. Education for caregivers of infants with single ventricle disease include guidelines to call health care providers (HCPs) in cases of hemodynamic interstage concerns, and symptom management questions, based on home monitoring of oxygen saturation and weight gain. There are variations in the staffing structure between pediatric hospitals but the programs often include care coordination and education by a nurse or advanced practice nurse communicating with parents in a reactive model waiting for data to be reported.

mHealth is defined through the National Institutes of Health (NIH) as the use of mobile and wireless devices to improve health outcomes, service, and research. The use of applications is widespread in adult care with estimated 40,000 health-care applications available. Some studies in pediatric medical homes have shown association of mHealth with adherence and self-monitoring to improved outcomes. mHealth innovations like the Cardiac High Acuity Monitoring Program (CHAMP) and other applications work most effectively when caregivers and interstage programs work together to improve care and are a focus of future research from the National Institute of Nursing Research. Much of the recent interstage literature focuses on mortality and weight measures with little focus on expanding types of outcomes to the parental and interstage teams' perspectives and phenomena like infant development.

Recent developments in technology can provide a proactive means for data transfer for home symptom monitoring so the interstage nursing team can review trends and provide proactive monitoring for infants in the interstage. Since 2012, two pilot studies have been published illustrating varying types of mHealth for the interstage with outcomes of improved somatic growth and an improved system of interstage data review but did not show significant mortality improvements. An innovative mHealth technology, CHAMP, was begun in 2014 for interstage home monitoring symptom management and found improved interstage mortality outcomes compared with historical controls. Research gaps remain in the role of adherence in this population to the mHealth technology and the parental experience of utilizing these innovative methods for communication with the clinical team.

Rationale The purpose of this study is to provide a rich description of the parental perspectives of utilizing a mHealth application for data transfer during the single ventricle interstage monitoring period for infants with congenital heart disease. The use of the case study design in healthcare has been encouraged by Robert Yin because it adapts to the complexity of interactions in a system that may be rapidly changing. Yin's qualitative case research "design propositions", presented below for this study, are applied to the literature and the PI's professional experience to focus the scope of the study and improve feasibility of completion of this qualitative case study approach research study. Propositions in this type of qualitative design are similar to hypothesis in quantitative designs to help formulate themes emerging from the data. The use of propositions may help with contributions for the body of knowledge after generalizing case study analysis, especially in cases of critical or extreme cases. Comparative analysis of the theoretical target (non-adherent parents) and rival cases (adherent parents) within the case study are improved with study propositions to guide the organization of data.

Study Propositions:

1. The parental perspectives of the interstage period will influence the use of a home monitoring mHealth technology
2. Parental perception of non-adherence of CHAMP and communication to the clinical team will match the actual non-adherence patterns of the mHealth innovation
3. The use of Cardiac High Acuity Monitoring Program (CHAMP) application from the parental perspective will benefit future improvements in this technology
4. Parents of infants with single ventricle will report the interstage report as a stressful time

Research Design

Methods. The proposed research study uses a comparative case study methodology, utilizing multiple sources of data to deeply examine 8-10 "cases," each of which is defined as parent(s) of a child (< 5 years of age) with single ventricle disease who used the mHealth application. One group of cases (4-5) will have used the mHealth application less than recommended (non-adherent to the home monitoring recommendations) or declined to use the application and returned it before the end of the interstage period. The other group of comparison cases (4-5 cases) will have used the application as recommended by the clinical team (adherent) and continued doing so through the interstage period.

Yin defines various types of cases, including, explanatory or causal case studies, descriptive case studies, and exploratory case studies. The cases in this study are exploratory in that they focus on "what" can be learned from these cases of using a novel mHealth innovation and the CHAMP care team as a unit. Across the U.S., nearly 2,000 infants are born with single ventricle cardiac disease each year but the actual experience at home is difficult to comprehend. The research design is a multiple case study design with embedded units of non-adherent and adherent cases of parental use of CHAMP within the larger case group through the CHAMP Clinic at Children's Mercy Kansas City.

Data sources will include semi-structured interviews with parents that include observations of simulated home monitoring equipment and processes that had been previously used including location, time of day, and frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Adult over 18 years of age parent(s) of children with single ventricle cardiac disease
2. Parent(s) of children were discharge home in the interstage period from December 2013 to May 2017 that have completed the interstage period with Stage II Glenn cardiac surgery as of June 8th, 2017.
3. Parents(s) of children who were followed in the CHAMP clinic at Children's Mercy.
4. Parent(s) of CHAMP children who had the CHAMP mHealth application (CHAMP App) available for transfer of home monitoring data during the interstage

Exclusion Criteria:

1. Non-English speaking parent(s)
2. Parent(s) of children who were not discharged interstage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Purposeful sampling will be used for recruiting among the first 80 infants from that used Cardiac High Acuity Monitoring Program (CHAMP) mHealth. All single and dual parent case sets will be recruited from a single tertiary center's pediatric cardiology department that used a mHealth application during the interstage period with the single ventricle team clinic known as CHAMP. Thus a case will be defined as the parent(s) of a single ventricle child who utilized CHAMP to monitor their baby at home during interstage with preliminary screening from the CHAMP Webportal through Children's Mercy Kansas City.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Adherence to technology | 6 months
  parental perspective on interstage period will influence the number of Data days during the interstage period

SECONDARY OUTCOMES:
Non-adherence to mHealth technology | 6 months
  Parental perception of non-adherence of mHealth (CHAMP) and communication to the clinical team will match the actual non-adherence patterns of the mHealth innovation
Parental Stress | 6 months
  Parents of infants with single ventricle will report the interstage report as a stressful time

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, MSN, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shirali G, Erickson L, Apperson J, Goggin K, Williams D, Reid K, Bradley-Ewing A, Tucker D, Bingler M, Spertus J, Rabbitt L, Stroup R. Harnessing Teams and Technology to Improve Outcomes in Infants With Single Ventricle. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):303-11. doi: 10.1161/CIRCOUTCOMES.115.002452. Epub 2016 May 10. PMID 27166202
- [Background] Yin RK. Enhancing the quality of case studies in health services research. Health Serv Res. 1999 Dec;34(5 Pt 2):1209-24. PMID 10591280
- [Background] Black AK, Sadanala UK, Mascio CE, Hornung CA, Keller BB. Challenges in implementing a pediatric cardiovascular home telehealth project. Telemed J E Health. 2014 Sep;20(9):858-67. doi: 10.1089/tmj.2013.0343. Epub 2014 Aug 1. PMID 25083905
- [Background] Rempel GR, Harrison MJ. Safeguarding precarious survival: parenting children who have life-threatening heart disease. Qual Health Res. 2007 Jul;17(6):824-37. doi: 10.1177/1049732307303164. PMID 17582024